CLINICAL TRIAL: NCT01638936
Title: A Phase I/IIa Multi-dose Escalation Study of BT062 in Combination With Lenalidomide or Pomalidomide and Dexamethasone in Subjects With Relapsed or Relapsed/Refractory Multiple Myeloma
Brief Title: BT062 in Combination With Lenalidomide or Pomalidomide and Dexamethasone in Patients With Multiple Myeloma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Biotest Pharmaceuticals Corporation (Industry)
Collaborators: Biotest (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 983
Record Dates: First submitted 2012-03-08; First posted 2012-07-12 (Estimated); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Multiple Myeloma
Keywords: Combination; Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Administration, Intravenous; indatuximab ravtansine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- BT062 (Experimental): BT062 administered intravenously on days 1, 8 and 15 of each 28-day cycle, and lenalidomide or pomalidomide and dexamethasone administered orally to subjects with relapsed or relapsed/refractory MM
  Interventions: Drug: BT062 , intravenous administration

INTERVENTIONS:
Drug: BT062 , intravenous administration — Dose escalation to determine dose limiting toxicities (DLTs) and/or the maximum tolerated dose (MTD)/recommended Phase II dose (RPTD) of BT062 in combination with lenalidomide/dexamethasone
  Other Names: Indatuximab Ravtansine

SUMMARY:
The purpose of this study is to test safety and anti-tumor activity of BT062 in combination with lenalidomide and dexamethasone to define the best doses for treating patients with relapsed and refractory multiple myeloma.

DETAILED DESCRIPTION:
BT062 is an antibody-drug conjugate designed to bind and destroy Myeloma cells. The study drug is being given in multiple doses with standard Multiple Myeloma treatments, lenalidomide and dexamethasone, to test how well the treatments are tolerated and work together. This study is a dose escalation study with the purpose to find out the highest dose of BT062 that a subject can tolerate in combination with lenalidomide and dexamethasone.

ELIGIBILITY:
Inclusion Criteria

* Diagnosis of active Multiple Myeloma according to the International Myeloma Working Group (IMWG) diagnostic criteria
* Relapsed or relapsed/refractory progressive Multiple Myeloma
* Subjects who failed at least one prior therapy (BT062/Len/dex)
* Subjects who failed at least two prior therapy (BT062/Pom/dex)
* Subjects age ≥18 years
* Life expectancy of ≥12 weeks
* Eastern Cooperative Oncology Group (ECOG) performance status (Zubrod) ≤2
* Normal organ and bone marrow
* Signed written informed consent in accordance with federal, local, and institutional guidelines
* Subjects must agree to follow all Guidelines from REVLIMID REMS Program or POMALYST REMS
* Women of child bearing potential (WCBP), must agree to use 2 contraceptive methods

Exclusion Criteria:

* Chemotherapy or radiotherapy within 3 weeks (6 weeks for nitrosoureas or mitomycin C) prior to day 1 or those who have not recovered from adverse events (AEs) due to agents administered more than 3 weeks earlier
* Antineoplastic therapy with biological agents within 2 weeks before day 1 or within 5 drug half-lives (t½) prior to first dose, whichever time period is longer
* Concomitant antineoplastic therapies including chemotherapy, radiotherapy, or biological agents during the study
* Treatment with another investigational drug during the study or within 3 weeks before day 1 or within 5 drug half-live (t½) prior to first dose, whichever time period is longer
* Treatment with BT062 in previous studies
* Major surgery within 4 weeks before day 1 (this does not include placement of vascular access device or tumor biopsies)
* Malignancy within 3 years before day 1, other than the trial indication multiple myeloma and excluding treated non-melanoma skin cancer, superficial bladder cancer, carcinoma in-situ of the cervix and prostate carcinoma ≤ Gleason Grade 6 with stable prostate specific antigen (PSA) levels
* Subjects with plasma cell leukemia (PCL)
* Subjects with deep vein thrombosis (DVT) and Pulmonary embolism (PE) within 3 months prior to day 1 treatment
* Severe infections necessitating use of antibiotics / antivirals during the screening period
* Clinically relevant active infection including active hepatitis B or C or human immunodeficiency virus (HBV, HCV, or HIV) or any other concurrent disease
* Acute or relevant abnormalities in electrocardiogram (ECG)
* Significant cardiac disease
* Pregnant or breast-feeding
* Positive serum or urine pregnancy test
* Hypersensitivity to the active substance or to any of the excipients for study drug BT062, or history of severe allergic or anaphylactic reaction to therapeutic proteins (e.g. reaction to vaccination or to biological therapy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2012-07-03 (Actual); Primary Completion 2018-10-30 (Actual); Study Completion 2018-10-30 (Actual)

PRIMARY OUTCOMES:
Determination of optimal dose of BT062 (Phase I part) | 6 months
  The Phase I part will follow a standard dose escalation design with at least 3 patients per dose level to define optimal dose of BT062 in combination with lenalidomide/dexamethasone. Optimal dose will be defined by dose limiting toxicities (DLT) observed during Cycle 1 (28 days).
Evaluation of response (Phase IIa part) | 18 months
  Response to treatment with optimal dose of BT062 (defined in Phase I part) in combination with lenalidomide/dexamethasone or pomalidomide/dexamethasone will be evaluated at baseline and at start of each Cycle (every 28 days). Response evaluation will be primarily based on assessment of M-protein and serum free light chains. If clinically required bone marrow analysis, plasmacytoma evaluation, and skeletal survey will be performed.

SECONDARY OUTCOMES:
Qualitative toxicities of BT062 in combination with lenalidomide/dexamethasone or pomalidomide/dexamethasone | 24 months
  Safety will be assessed at each visit by incidence of adverse events and by clinically significant changes in the patients physical examination, vital signs, and clinically laboratory results
Pharmacokinetics of BT062 in combination with lenalidomide/dexamethasone or pomalidomide/dexamethasone | 24 months
  Pharmacokinetic parameters will be assessed from plasma by measuring intact BT062 and free maytansinoid (DM4)
Assessment of Time To Event end points | 24 months
  Based on the response evaluation, the following Time To Event end points will be evaluated: Time To Progression, Progression Free Survival, Time To Next Treatment, Duration Of Response, Overall survival.
Quantitative toxicities of BT062 in combination with lenalidomide/dexamethasone or pomalidomide/dexamethasone | 24 months
  Safety will be assessed at each visit by incidence of adverse events and by clinically significant changes in the patients physical examination, vital signs, and clinically laboratory results

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth C Anderson, MD, Study Director — Dana-Farber Cancer Institute
Locations (10):
- United States (10):
  - City of Hope, Duarte, California
  - USC Norris Comprehensive Cancer Center, Los Angeles, California
  - Mayo Clinic, Jacksonville, Florida
  - Memorial Healthcare System, Pembroke Pines, Florida
  - Emory University Winship Cancer Institute, Atlanta, Georgia
  - The University of Chicago, Chicago, Illinois
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Mount Sinai Medical Center, New York, New York
  - University of Texas Health Science Center, San Antonio, Texas

REFERENCES:
- [Derived] Kelly KR, Ailawadhi S, Siegel DS, Heffner LT, Somlo G, Jagannath S, Zimmerman TM, Munshi NC, Madan S, Chanan-Khan A, Lonial S, Chandwani S, Minasyan A, Ruehle M, Barmaki-Rad F, Abdolzade-Bavil A, Rharbaoui F, Herrmann-Keiner E, Haeder T, Wartenberg-Demand A, Anderson KC. Indatuximab ravtansine plus dexamethasone with lenalidomide or pomalidomide in relapsed or refractory multiple myeloma: a multicentre, phase 1/2a study. Lancet Haematol. 2021 Nov;8(11):e794-e807. doi: 10.1016/S2352-3026(21)00208-8. Epub 2021 Sep 13. PMID 34529955